CLINICAL TRIAL: NCT01191957
Title: Randomized Study Comparing i.v. Busulfan (Busilvex®) Plus Fludarabine (BuFlu) Versus Busilvex® Plus Cyclophosphamide (BuCy2) as Conditioning Regimens Prior AlloHSCT in Patients (Age >= 40 and =<65 Years) With AML in Complete Remission.
Brief Title: Busulfan (BU) Plus Fludarabine Vs Intravenous BU Plus Cyclophosphamide as Conditioning Regimens Prior Allogeneic Hematopoetic Stem Cells Transplant (HSCT) in AML
Acronym: GITMO-AMLR2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GITMO AMLR2
Record Dates: First submitted 2010-06-10; First posted 2010-08-31 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia; Allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Busulfan; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I. V. Busulphan plus Cyclophosphamide (Active Comparator): Conventional conditioning regimen with intravenous (i.v.) Busulphan (Busilvex), 12.8 mg/kg followed by Cyclophosphamide, 120 mg/kg iv.
  Interventions: Drug: Busulphan plus Cyclophosphamide
- I. V. Busulphan plus Fludarabine (Experimental): Reduced toxicity conditioning regimen with intravenous (i.v.)Busulphan (Busilvex), 12.8 mg/kg plus Fludarabine, 4 x 40 mg/m².
  Interventions: Drug: Busulphan plus Fludarabine

INTERVENTIONS:
Drug: Busulphan plus Cyclophosphamide — I.V. Bu (Busilvex), 12.8 mg/kg:
  Day -9: 0.8 mg/kg/dose x 4 doses Day -8: 0.8 mg/kg/dose x 4 doses Day -7: 0.8 mg/kg/dose x 4 doses Day -6: 0.8 mg/kg/dose x 4 doses Day -5: Rest
  Followed by:
  Cyclophosphamide, 120 mg/kg iv:
  Day -4: 60 mg/kg Day -3: 60 mg/kg
  Other Names: I.V. BuCy2
  Arms: I. V. Busulphan plus Cyclophosphamide
Drug: Busulphan plus Fludarabine — I.V. Bu (Busilvex), 12.8 mg/kg:
  Day -6: 0.8 mg/kg/dose x 4 doses Day -5: 0.8 mg/kg/dose x 4 doses Day -4: 0.8 mg/kg/dose x 4 doses Day -3: 0.8 mg/kg/dose x 4 doses plus:
  Fludarabine, 4 x 40 mg/m² iv:
  Day -6: 40 mg/m² Day -5: 40 mg/m² Day -4: 40 mg/m² Day -3: 40 mg/m²
  Other Names: I.V. BuFlu
  Arms: I. V. Busulphan plus Fludarabine

SUMMARY:
The purpose of this prospective phase III, open-label, randomized multicenter study is to evaluate whether Acute Myeloid Leukemia (AML) elderly patients in Complete Remission (CR) undergoing allogeneic hematopoietic stem cell transplantation after a reduce toxicity conditioning regimen (I.V. BuFlu) as compared to the conventional I.V.

BuCy2 program will experience:

1. A lower transplant-related mortality (TRM) at 1 year after Hematopoietic Stem Cells Transplant (HSCT)
2. A similar anti-leukemic activity and a similar or better safety profile, in terms of:

   * Early and/or late graft rejection
   * Hematopoietic and immunologic recovery
   * Chimerism
   * Toxicity and incidence of Veno-occlusive Disease (VOD)
   * Acute (aGvHD) and chronic graft-versus-host disease (cGvHD)
   * Cumulative incidence of TRM at +100 days and 2 years after transplant
   * Cumulative incidence of relapse by 1 and 2 years after transplant
   * Event-free (EFS) and overall survival (OS) by 1 and 2 years after transplant

DETAILED DESCRIPTION:
Hematopoietic stem-cell transplantation (HSCT) is a potentially curative treatment modality for patients with Acute Myelogenous Leukemia (AML).

An effective conditioning regimen is based on the association of oral Busulfan 4 mg/kg daily in 4 doses, each of 1 mg/kg, on each of 4 successive days (total dose, 16 mgkg), followed by CY 60 mg/kg intravenously on each of 2 successive days (BuCy2). The antileukemic activity of this latter program was tested and confirmed in most large randomized clinical trials conducted in AML and Chronic Myeloid Leukemia (CML) patients in which the BU-CY regimen was associated with survival and relapse probabilities that compare favourably with the CY-Total Body Irradiation (TBI) regimen. The BuCy2 program is considered a golden standard preparative regimen for allogeneic transplantation in AML patients.

Nonetheless, for many years the treatment related toxicities of all these full myeloablative conditioning regimens has substantially limited the overall applicability of the transplant procedure to young patients with a good performance status (PS). The observation that allogeneic stem cell transplants have a potentially curative graft-versus-leukemia (GVL) effect in addition to the antileukemic action of myeloablative conditioning regimens was a major stimulus for the development of reduced-intensity conditioning (RIC) regimens, aimed primarily at securing engraftment to provide the GVL effect, while minimizing regimen-related toxicity.

The observation that allogeneic stem cell transplants have a potentially curative graft-versus-leukemia (GVL) effect in addition to the antileukemic action of myeloablative conditioning regimens was a major stimulus for the development of reduced-intensity conditioning (RIC) regimens, aimed primarily at securing engraftment to provide the GVL effect, while minimizing regimen-related toxicity. As a consequence reduced-intensity conditioning (RIC) regimens might give possibility to extend access to allogeneic transplantation to patients who would not have previously been considered reasonable candidates because of their age and for the presence of comorbidities. However, after a lot of initial enthusiasm, it has become clear that a more intensive conditioning is associated with a reduced risk for relapse after HSCT. Therefore, while it is clear that RIC transplants have opened the way to using allogeneic SCT in patients several years older than the upper age limit of 60, the superiority of the RIC approach cannot be assumed even in this subgroup of patients. This is why, more recently, investigators are looking for conditioning programs that while better tolerated still might retain a strong ability of inducing a direct ablation of the leukemic hematopoiesis. This has led to the new concept of reduced toxicity rather than reduced intensity conditioning programs. One of such a program is based on the association of a myeloablative dose of intravenous Busulfan (0.8 mg/kg/d for 4 days), with Fludarabine (30 mg/m2/d for 4 days) which has been reported as highly effective in patients with AML. In elderly patients with this disease, this program might lead to an overall outcome at least as good as that following conventional myeloablative programs such as those based on Cyclophosphamide combined to the same dose of IV Busulfan or the TBI. In fact, when compared to these latter programs, the Busulfan Fludarabine regimen was found associated with lower non relapse mortality although a higher relapse rate was still documented, but not in all published experiences. In all, outcomes for standard transplant regimens have generally improved and these newer myeloablative regimens of Fludarabine with full-dose intravenous Busulfan achieve 1 year TRM below 10%. So, based on these considerations, protocol GITMO-AML.R2 has been designed to compare intravenous Busulfan plus Fludarabine (BuFlu) versus Busulfan (I.V. Bu; Busilvex®) plus Cyclophosphamide (BuCy2) as conditioning regimens prior to allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT) in patients (aged between 40 and 65 years) with Acute Myeloid Leukemia (AML) in Complete Remission (CR).

So, based on these considerations, protocol GITMO-AML.R2 has been designed to compare intravenous Busulfan plus Fludarabine (BuFlu) versus Busulfan (I.V. Bu; Busilvex®) plus Cyclophosphamide (BuCy2) as conditioning regimens prior to allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT) in patients (aged between 40 and 65 years) with Acute Myeloid Leukemia (AML) in Complete Remission (CR).

The principal objective of this trial is the evaluation of one year transplant-related mortality (TRM) of AML patients undergoing allogeneic hematopoietic stem cell transplantation after a reduced toxicity conditioning regimen (I.V.BuFlu) as compared to the conventional I.V. BuCy2 program.

To this purpose, in the IV BuCy2 arm, reference TRM was assumed to be 25% (range 16-50%) while in the IV BuFlu arm and an estimated 12.5% TRM is assumed (range 0-30%). The study is designed to demonstrate a relative risk reduction of 50%. For the event-driven two-sided test, an alpha-level probability of 0.05 (type I error) and a power of 80% (type II error=0.2) has been considered. The ratio between the numbers of patients included in each arm is set equal to 1:1. The resulting required sample size is 240 (120 patients in each arm). Sample size estimation is based on the intention-to-treat principle.

The accrual time is 2.5 years, and an additional follow-up of 2 years is planned after the last patient entry in the study and before the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients
* Age more than 40 and less than 65 years
* Diagnosis of AML (FAB or WHO classification) in Complete Remission (CR)
* Availability of an HLA compatible sibling or unrelated donor
* Performance status : Eastern Cooperative Oncology Group (ECOG)<3
* Written and signed informed consent
* Central Venous access (Central KT) secured through an indwelling catheter.
* Life expectancy not severely limited by concomitant illness. Donors
* Age between 18 years and 65 years inclusive.
* Availability of an HLA-identical sibling donor (MRD) or HLA-compatible unrelated donor (MUD). Donor selection is based on molecular high-resolution typing (4 digits) of the HLA gene loci class I (HLA- A, B, and C) and class II (DRB1). In case, no class I and class II completely identical donor (8 out of 8 gene loci) can be identified, one antigen/allele disparity (class I) or one allele disparity (class II, DRB1) between patient and donor are acceptable. In any cases the degree of histocompatibility between patient and donor must fulfill with the minimal degree of matching established by the Italian Bone Marrow Donor Registry.

Exclusion Criteria:

Patients

* AML patients in 1st CR with:

  * t(15;17) or promyelocytic leukemia/retinoic acid receptor gene translocation, PML/RARα positive APL
  * t(8;21)(q22;q22) with white blood cells (WBC) count at diagnosis less than 20 x 109/L without additional adverse cytogenetic abnormalities.
  * inv(16) or t(16;16)(p13;q22) without additional adverse cytogenetic abnormalities.
* Previous allogeneic transplantation Poorly controlled arterial hypertension with blood pressure above 150/90 on standard medication
* Acute Myocardial Infarction (AMI) within the last 12 months
* Positive pregnancy test (in women not in menopause)
* Positive HIV serology
* Any major organ dysfunction
* Pulmonary dysfunction (Fraction Ejection Volume, FEV1 <40%, Diffusing Capacity of Lung for carbon monoxide, DLCO <50%,)
* Hepatic dysfunction (Serum bilirubin >1.5 mg% or serum transaminases >2x UNL)
* Chronic active hepatitis or cirrhosis
* Cardiac dysfunction (LVEF <40)
* Chronic renal insufficiency (Serum creatinine >1.5 mg/dl or creatinine clearance <=50 ml/min)
* Invasive fungal infection still evolutive at the time of registration
* Central nervous system involvement
* Uncontrolled oral/dental infections
* Abnormal dental evaluation
* Patient has another progressive malignant disease or a history of other malignancies within 2 years prior to study entry
* Severe psychiatric illness or any disorder that compromises ability to give truly informed consent for participation in this study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
transplant-related mortality (TRM) | 1 year post transplant
  The primary endpoint is to determine the cumulative incidence of transplant related mortality (TRM) defined as non-relapse mortality. Assessment will be performed at 1 year after transplantation.
  TRM will be defined as any death by causes other than relapse and/or progressive disease. Deaths after persistent post-transplant relapse will be categorized as due to the disease irrespective of the proximate cause.

SECONDARY OUTCOMES:
Assessment in the two arms of the safety and efficacy profile | 30-60-100-180 days, 1-2 years
  Assessment in the two arms of the safety and efficacy profile defined as: early and/or late graft rejection, hematopoietic recovery, chimerism, toxicity and incidence of VOD, incidence and severity of acute (aGvHD) and chronic graft-versus-host disease (cGvHD), cumulative incidence of TRM, relapse, event-free (EFS) and overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro AR Rambaldi, Professor, Principal Investigator — A.O. Papa Giovanni XXIII
Locations (26):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Italy (25):
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera SS Antonio e Biagio, Alessandria
  - Clinica di Ematologia - Ospedali Riuniti di Ancona, Ancona
  - Policlinico di Bari-Ematologia con trapianti, Bari
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale Regionale Generale- Divisione Ematologia, Bolzano
  - AO Spedali Civili di Brescia- USD - TMO Adulti, Brescia
  - Ospedale Ferrarotto - Ematologia, Catania
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Cattedra di Ematologia - Azienda Ospedaliera di Careggi, Florence
  - AOU-IRCCS San Martino-IST Ematologia II, Genova
  - Divisione di Ematologia - Istituto Nazionale dei Tumori, Milan
  - U.O. Ematologia I - Centro Trapianti di Midollo - Ospedale Maggiore - Policlinico Mangiagalli e Regina Elena, Milan
  - Cattedra di Medicina Interna ed Ematologia - Ospedale S. Gerardo de' i Tintori - Università degli Studi di Milano, Monza
  - A.O.U. Policlinico Federico II, Napoli
  - AOR Villa Sofia-Cervello - Bone Marrow Transplant Unit, Palermo
  - IRCCS Policlinico S. Matteo, Pavia
  - Dip. di Ematologia - Unità di Terapia Intensiva Ematologica per il Trapianto Emopoietico - Ospedale Civile di Pescara, Pescara
  - Divisione di Ematologia - Istituto di Semeiotica Medica - Policlinico A. Gemelli, Roma
  - Policlinico Universitario Tor Vergata, Roma
  - Sapienza University, Roma
  - Az. Ospedaliera Universitaria Senese - Divisione Ematologia e Trapianti, Siena
  - AOU Città della Salute e della Scienza, Torino
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Ospedale S. Bortolo-Divisione Ematologia, Vicenza

REFERENCES:
- [Derived] Rambaldi A, Grassi A, Masciulli A, Boschini C, Mico MC, Busca A, Bruno B, Cavattoni I, Santarone S, Raimondi R, Montanari M, Milone G, Chiusolo P, Pastore D, Guidi S, Patriarca F, Risitano AM, Saporiti G, Pini M, Terruzzi E, Arcese W, Marotta G, Carella AM, Nagler A, Russo D, Corradini P, Alessandrino EP, Torelli GF, Scime R, Mordini N, Oldani E, Marfisi RM, Bacigalupo A, Bosi A. Busulfan plus cyclophosphamide versus busulfan plus fludarabine as a preparative regimen for allogeneic haemopoietic stem-cell transplantation in patients with acute myeloid leukaemia: an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2015 Nov;16(15):1525-1536. doi: 10.1016/S1470-2045(15)00200-4. Epub 2015 Sep 28. PMID 26429297